CLINICAL TRIAL: NCT05941143
Title: Effect of Mindfulness on EEG Brain Activity for Cognitive and Psychological Well-being in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro San Giovanni di Dio Fatebenefratelli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 104/18
Record Dates: First submitted 2023-06-16; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-06

CONDITIONS: Healthy Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mindfulness-based intervention (Experimental): The intervention consist of 8 sessions in which participants learned three main different practices: body scan, sitting meditation, and yoga practice. Participants are instructed to regularly engage in home mindfulness practice of these new learned skills (45 minutes a day for 6 days a week). Home exercises include formal mindfulness practice (i.e., meditation and yoga) for about 30-35 minutes a day and informal practice focused on bringing mindful awareness to everyday activities for about 10-15 minutes a day. Mp3 audio of meditations proposed at each session are provided to guide personal practice.
  Interventions: Other: mindfulness-based intervention

INTERVENTIONS:
Other: mindfulness-based intervention — 8 weekly group 2-hour sessions program adapted from mindfulness-based stress reduction and mindfulness-based cognitive therapy protocols. It was specifically tailored to older adults.

SUMMARY:
As the worldwide population of older adults rapidly increases over the coming years, effective strategies are needed to help this population to maintain and enhance physical, cognitive, and psychological well-being. Up to 10% of community dwelling older adults have depressive symptoms in Europe. Older adults are also subject to chronic illnesses which further exacerbate psychological symptoms. Furthermore, normal aging is associated with decline in cognitive functioning. Given the prevalence of mental health problems and cognitive difficulties in older adults, mindfulness-based interventions (MBIs) could be helpful in this population. Accordingly, a growing number of studies suggest that mindfulness-based interventions in the elderly have beneficial effects on psychological health (decrease in depression, anxiety, sleep problems, and increase in general mood and positive affect) and cognition (enhanced attention, executive functions).

Electroencephalography (EEG) is a non-invasive technique which can be useful to study the neurophysiological correlates of mindfulness, and give neurobiological evidence of its beneficial effect in the elderly. Studies that examined spectral power outcomes between mindfulness and control state showed (i) increased alpha and theta power, as a marker of internally-directed attention processing and executive functioning and (ii) a shift towards left-sided anterior alpha activation, a pattern associated previously with positive emotions.

The aim of this study is to evaluate short and long-term cognitive, psychological, and physiological effects of a standard 8-week MBI in healthy older adults. Cognitive and psychological evaluations, and resting state EEG will be administered within 2 weeks prior to and within 2 weeks following MBI, and repeated 24 weeks following MBI.

DETAILED DESCRIPTION:
Sixty older adults will be enrolled through local media announcements, meetings with elderly people organized in collaboration with local leisure and cultural associations, Alzheimer cafè, university of the third age, contacts with general practitioners. All participants will undergo cognitive and psychological evaluation and EEG. Moreover, current pharmacological therapies will be recorded and medical illness burden and comorbidity will be rated by the Cumulative Illness Rating Scale. Personality traits will be assessed by the Revised NEO Personality Inventory (NEO PI-R). The Subjective Cognitive Decline-Interview will be administered to evaluate the presence of subjective cognitive decline.

The EEG will be recorded (250 Hz sampling frequency, without filtering) with 19 standard electrodes positioned according to the international standard 10-20 in baseline conditions. The electrodes will have an impedance of less than 5 kiloohm. Recordings of 5 minutes with open eyes and 5 minutes with eyes closed will be performed. Following the acquisition of the signal, spectral analysis will be applied.

Mindfulness-based intervention is a standardized program which consists of 2-hour sessions that will be delivered at weekly intervals for 8 weeks in group setting. It is based on a comprehensive set of mindfulness practices derived from mindfulness-based stress reduction and mindfulness-based cognitive therapy programs, but specifically tailored to older adults. Participants will also be instructed to regularly engage in home mindfulness practice.

Follow-up: all participants will repeat cognitive and psychological evaluation and EEG after 2 weeks and after 24 weeks from the end of MBI.

Data analysis: Descriptive statistics on cognitive, psychological, and EEG variables will be done by using parametric and non- parametric tests. The analyses of correlation between different clinical variables (assessment tools) and EEG brain features will be assessed by linear and generalized linear models. For longitudinal analyses we will adopt the generalized estimating equation models.

ELIGIBILITY:
Inclusion criteria:

* community-dwelling older adults
* age between 60 and 75 years
* normal cognition

Exclusion criteria:

* clinically significant depression or anxiety
* major neurological disorders (i.e., stroke, dementia or cognitive impairment, tumor)
* major psychiatric disorders (i.e., major depressive disorder, bipolar disorder, drug and alcohol dependence)
* chronic disease or acute unstable illness (respiratory, cardiovascular, digestive, renal, metabolic, hematologic, endocrine, infectious, or malignancy) which interfered with the aims of the study protocol.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline in dispositional mindfulness on the Five Facet Mindfulness (FFM) Scale at week 8 | week 8
  FFM scale is a validated self-reported scale assessing dispositional mindfulness, with higher scores indicating higher mindfulness. Change=8 week score-baseline score.
Change from baseline in verbal memory on the California Verbal Learning Test (CVLT) at week 8 | week 8
  CVLT is a validated word-list task assessing verbal memory, with higher scores indicating better verbal memory. Change=week 8 score-baseline score.
Change from baseline in interoceptive mindfulness on the Multidimensional Assessment of Interoceptive Awareness (MAIA) scale at week 8 | week 8
  MAIA is a 32-item validated self-reported scale assessing interoceptive awareness, with higher scores indicating higher awareness. Change=8 week score-baseline score.

SECONDARY OUTCOMES:
Change from baseline EEG alpha power at week 8 | week 8
  alpha 1, alpha 2, alpha 3 bands

OTHER OUTCOMES:
Change from baseline in emotion regulation strategies on the Emotion Regulation Questionnaire (ERQ) scale at week 8 | week 8
  ERQ scale is a validated self-reported scale assessing emotion regulation strategies, with higher scores indicating better emotion regulation. Change=week 8 score-baseline score.
Change from baseline in emotion regulation strategies on the Heidelberg Form for Emotion Regulation Strategies (HFERST) scale at week 8 | week 8
  HFERST is a validated self-reported scale assessing emotion regulation strategies, with higher scores indicating a more frequent use of the strategies. Change=week 8 score-baseline score.
Change from baseline in chronic worry on the Penn State Worry Questionnaire (PSWQ) at week 8 | week 8
  PSWQ is a validated self-reported scale assessing chronic worry, with higher scores indicating higher worries. Change=week 8 score-baseline score.
Change from baseline in psychological well-being on the Warwick-Edinburgh Mental Well-being scale at week 8 | week 8
  Warwick-Edinburgh Mental Well-being is a validated self-reported scale assessing psychological well-being, with higher scores indicating higher well-being. Change=week 8 score-baseline score.
Change from baseline in attention function on the Attentional Matrices test at week 8 | week 8
  Attentional Matrices is a validated objective test assessing attention, with higher scores indicating better attention. Change=week 8 score-baseline score.
Change from baseline in attention function on the Trail Making Test A (TMTA) at week 8 | week 8
  TMTA is a validated objective test assessing attention, with lower scores indicating better attention. Change=week 8 score-baseline score.
Change from baseline in executive functions on the Wisconsin Card Sorting Test (WCST) at week 8 | week 8
  WCST is a validated objective test assessing cognitive flexibility, with lower scores indicating better function. Change=week 8 score-baseline score.
Change from baseline in executive functions on the Stroop test at week 8 | week 8
  Stroop test is a validated objective test assessing the effects of interference on reading ability, with higher scores indicating better performance and less interference on reading ability. Change=week 8 score-baseline score.
Change from baseline in executive functions on Trail Making Test B (TMTB) at week 8 | week 8
  TMTB is a validated objective test assessing executive functions, with lower scores indicating better function. Change=week 8 score-baseline score.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Centro San Giovanni di Dio Fatebenefratelli, Brescia, Italy

IPD SHARING:
Plan to Share IPD: Yes
The dataset analyzed in this article is publicly available at the Mendeley data repository
Supporting Information: Analytic Code
URL: https://data.mendeley.com/datasets/x3vb85t4xh/1

REFERENCES:
- [Derived] Galluzzi S, Lanfredi M, Moretti DV, Rossi R, Meloni S, Tomasoni E, Frisoni GB, Chiesa A, Pievani M. Cognitive, psychological, and physiological effects of a web-based mindfulness intervention in older adults during the COVID-19 pandemic: an open study. BMC Geriatr. 2024 Feb 14;24(1):151. doi: 10.1186/s12877-024-04766-z. PMID 38350854